CLINICAL TRIAL: NCT05988411
Title: Ultrasound-Based Renal Sympathetic Denervation as Adjunctive Upstream Therapy During Atrial Fibrillation - Redo Ablation Procedures: A Pilot Study
Brief Title: ULTRA-HFIB-Redo: Ultrasound-based Renal Sympathetic Denervation vs Control in Redo Ablation Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vivek Reddy (Other)
Responsible Party: Sponsor-Investigator, Vivek Reddy, Professor of Medicine , Director, Cardiac Electrophysiology, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRANY 23-02-344
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Intervention Model Description: Prospective, controlled, single-blind, randomized (2:1, Intervention:Control) clinical trial.
Who Masked: Participant
Masking Description: single-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Catheter ablation + renal denervation (Experimental): Catheter ablation + renal denervation
  Interventions: Device: Renal Denervation; Device: Catheter Ablation
- Catheter ablation only (Active Comparator): Catheter ablation
  Interventions: Device: Catheter Ablation

INTERVENTIONS:
Device: Renal Denervation — Renal denervation using the Paradise renal denervation system - a dedicated Renal Denervation (RDN) catheter that delivers a circumferential ring of ablative ultrasound energy
  Arms: Catheter ablation + renal denervation
Device: Catheter Ablation — Catheter ablation - one of the most common procedures performed by Cardiac Electrophysiologists for atrial fibrillation.

SUMMARY:
This is a Prospective, controlled, single-blind, randomized (2:1, Intervention:Control) clinical trial. The purpose of the study is to determine the role of adjunctive renal sympathetic denervation in the prevention of Atrial Fibrillation (AF) recurrence in patients with hypertension scheduled for a redo AF ablation procedure for paroxysmal or persistent AF. Patients will be randomized to either i) AF ablation (Control) or ii) AF ablation + renal sympathetic denervation (Intervention).

DETAILED DESCRIPTION:
This is a prospective, controlled, single-blind, randomized trial. The pilot study will be conducted in up to 20 clinical sites in the United States. Once the clinical sites are up and running (expected to take 6 months), accrual is expected to take an additional 9 months, and all patients will be followed for 12 months post randomization. Patients, the Clinical Events Committee and the ECG core lab will be blinded during the trial. Patients will be unblinded at the 12-month visit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18;
* Planned for a redo AF ablation procedure (paroxysmal or persistent); (prior to randomization, a technically successful AF ablation procedure, defined as successful pulmonary vein isolation, if needed, as well as bidirectional block of any attempted anatomic lesion sets such as cavotricuspid isthmus line, roofline, mitral line and superior vena cava isolation, must have been completed). Note: the clinical recurrences must primarily be atrial fibrillation, and not atrial flutter/tachycardia (that is, a prospective patient may have a AFL/AT recurrences, but AF must be the dominant recurrent rhythm.)
* History of hypertension and either:

  * Documented history of SBP≥160 or DBP≥100, or;
  * Receiving ≥1 antihypertensive medication;
* Willingness to adhere to study restrictions and comply with all post-procedural follow-up requirements

Exclusion Criteria:

* Long-standing persistent AF (>12 months); >3 prior atrial fibrillation ablations (lifetime); AF ablation within 3 months of enrollment; extensive scar in left atrium.
* Individual with valvular AF or AF due to a reversible cause
* Prior treatment with other devices for hypertension including but not limited to ROX Coupler, Mobius stent, and/or the CVRx barostimulator device.
* NYHA class IV congestive heart failure;
* Individual has renal artery anatomy that is ineligible for treatment (as determined by renal angiography);

  * Main renal artery diameter <3mm or >8.0 mm
  * Main renal treatable artery length < 20 mm (length may include proximal branches)
  * Presence of renal artery stenosis of any origin ≥30%
  * Calcification in renal arteries
  * Prior renal denervation procedure
  * Presence of abnormal kidney tumors
  * Renal artery aneurysm
  * Pre-existing renal stent or history of renal artery angioplasty
  * Pre-existing aortic stent or history of aortic aneurysm
  * Fibromuscular disease of the renal arteries
  * Iliac/femoral artery stenosis precluding insertion of the Paradise Catheter
* Individual has an estimated glomerular filtration rate (eGFR) of less than 40mL/min/1.73m2, using the MDRD calculation;
* Inability to undergo AF catheter ablation (e.g., presence of a left atrial thrombus, contraindication to all anticoagulation)
* Individual with known allergy to contrast medium not amendable to treatment.
* Life expectancy <1 year for any medical condition
* Individual has experienced a myocardial infarction, unstable angina, cerebrovascular accident, or heart failure admission within 3 months of the baseline visit.
* Documented history of chronic active inflammatory bowel disorders such as Crohn's disease or ulcerative colitis.
* Female participants who are pregnant or nursing.
* Individual has known secondary hypertension.
* Individual has a single functioning kidney (either congenitally or iatrogenically).
* Individual has a known, unresolved history of drug use or alcohol dependency, lacks the ability to comprehend or follow instructions, or would be unlikely or unable to comply with study follow-up requirements.
* Patients concurrently enrolled in any other investigational drug or device trial that would interfere with the conduction of this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Freedom from atrial arrhythmias with no AADs | after 90 days
  Freedom from atrial arrhythmias (AT/AF/AFL) recurrence ≥ 30 seconds off all antiarrhythmic drug uses (AADs) (after the 90-day blanking period).

SECONDARY OUTCOMES:
Freedom from atrial arrhythmias (AT/AF/AFL) with AADs | at 12 months
  Freedom from AT/AF/AFL recurrence ≥ 30 seconds at 12 months (not including a 3-month blanking period) despite taking AADs
Procedure-related adverse events | at 12 months
  Number of procedure-related adverse events
Atrial Fibrillation Effect on Qualify of Life Questionnaire (AFEQT) | at 12 months
  Atrial Fibrillation Effect on Qualify of Life Questionnaire (AFEQT). Each item scored from 1-7, with total scale from 20-140, Lower score indicates better health outcomes.
Blood pressure | at 12 months
  Blood pressure - Systolic and Diastolic
Number of AF episodes | at 12 months
  AF burden assessed by the amount of AF episodes detected during Event Monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (8):
- United States (8):
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - UCSF, San Francisco, California
  - Los Robles Medical Center, Thousand Oaks, California
  - Henry Ford Health System, Detroit, Michigan
  - Mount Sinai Hospital, New York, New York
  - Trident Medical Center, Charleston, South Carolina
  - Christus, Tyler, Texas
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No